CLINICAL TRIAL: NCT02656602
Title: Computer-assisted Instruction Before Colonoscopy is as Effective as Nurse Counselling, a Controlled Trial (PAVO-E-EDUC)
Brief Title: Computer-assisted Instruction Before Colonoscopy is as Effective as Nurse Counselling, a Controlled Trial
Acronym: PAVO-E-EDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govert Veldhuijzen (Other)
Responsible Party: Sponsor-Investigator, Govert Veldhuijzen, Resident Gastroenterology, Medical Center Alkmaar
Organization: Medical Center Alkmaar (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: L013-011
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Colonoscopy; Education, Patient; eHealth
Keywords: Computer Assisted Instruction; Patient Counselling; Endoscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse Counseling (No Intervention): A trained endoscopy nurse provided patients with all information on their scheduled colonoscopy.
- Computer Assisted Instruction (Experimental): The computer assisted instruction consisted of a platform using video mimicking the patient journey with voice-over supported by photo's, 3D animation and instructive texts. The video was presented in short clips, maximal 45 seconds, to maintain the focus of patient. Patient interaction was ascertained by mandatory mouse-click after each item in the CAI.All elements of informed consent for colonoscopy (risks, alternatives) were included.
  Interventions: Other: Computer Assisted Instruction

INTERVENTIONS:
Other: Computer Assisted Instruction — The computer assisted instruction consisted of a platform using video mimicking the patient journey with voice-over supported by photo's, 3D animation and instructive texts. The video was presented in short clips, maximal 45 seconds, to maintain the focus of patient. Patient interaction was ascertained by mandatory mouse-click after each item in the CAI. All elements of informed consent for colonoscopy (risks, alternatives) were included.
  Other Names: MEx (Medical Experience)
  Arms: Computer Assisted Instruction

SUMMARY:
Better patient education prior to colonoscopy improves adherence to instructions for bowel preparation and leads to cleaner colons. The hypothesis of this trial is that computer assisted instruction (CAI) using video and 3D animations can maximize the effectiveness of nurse counselling and consequently improves bowel cleanliness. Furthermore, CAI will positively influence the patient experience.

Adults referred for colonoscopy were included in a Dutch large volume endoscopy unit. Exclusion criteria were illiteracy in Dutch and audiovisual handicaps. Patients were prospectively divided into two groups, one receiving nurse counselling and one receiving CAI and a nurse contact before colonoscopy. The main outcome, cleanliness of the colon during examination, was measured with the Ottawa Bowel Preparation Scale (OBPS) and the Boston Bowel Preparation Scale (BBPS). Patient comfort and anxiety were assessed at multiple time points: directly after the instruction and one hour before colonoscopy. Comfort was rescored 2 hours after colonoscopy. We also tested knowledge and comprehension one hour before colonoscopy. Statistical analyses included Mann-Whitney.

DETAILED DESCRIPTION:
To conduct the study, a prospective single center endoscopist blinded controlled design was used.

Patients Consecutive patients older than 18 years referred for elective colonoscopy were included from March 2013 until November 2013 in a single large volume endoscopy center (over 4000 colonoscopies/year) in the greater Amsterdam Area in the Netherlands. Exclusion criteria were illiteracy in Dutch and audiovisual/mental handicaps.

Study design After informed consent was obtained, patients were divided in two groups: the control group received nurse counselling and the intervention group received computer assisted instruction (CAI). Next, patients scored comfort ("How comfortable are you?") and patient anxiety ("How anxious are you)"on a 5-point Likert scale. (T1) After this, the CAI group had a contact with a trained endoscopy nurse for practical matters like bridging in anticoagulant therapy, insulin dosage calculation and scheduling of the colonoscopy. Next, patients were scheduled for their colonoscopies, maximum 6 weeks after the counselling session.

One hour prior to colonoscopy patients scored comfort and anxiety on the 5-point Likert scale. Also patient knowledge and comprehension was tested in a 10-question survey on the provided counselling information (T2).

Post-colonoscopy, patients re-scored comfort on the 5-point Likert scale (T3). During colonoscopy, the endoscopist assessed the bowel cleanliness with the Boston Bowel Preparation Scale (BBPS). For more subtle differences the Ottawa Bowel Preparation Scale (OBPS) was used.

Computer assisted instruction As intervention an interactive CAI was designed, according to current best practices, like good accessibility, plain language and engaging the user. Therefore the information was presented stepwise. The CAI consisted of a web-based platform using video mimicking the patient journey with voice-over supported by photo's, 3D animation and instructive texts. The video was presented in short clips, maximal 45 seconds, to maintain the focus of patient. Patient interaction was ascertained by mandatory mouse-click after each item in the CAI. All informative elements, especially mandatory for informed consent for colonoscopy (risks, alternatives) were included.

Outcomes The primary outcome was cleanliness of the colon during examination as assessed by the OBPS and the BBPS. The secondary outcomes were patient comfort, anxiety and knowledge and comprehension.

Statistical analyses The sample size of 350 provides 80% power, with a two-tailed α of 0.05, to detect an increase in the primary outcome measure from 6.0 in the control group to 6.3 in the experimental group.

All analyses were performed using SPSS version 20.0 for Windows (SPSS Inc., Chicago, IL, USA). Descriptive statistics were used to describe baseline information including frequency count, percentage and mean ±standard deviation. Further analyses included the chi-square test, independent t-test and Mann-Whitney. P-values under 0.05 were regarded statistically significant.

Ethical considerations The study was approved by the ethical and executive board of the institute.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years who were referred for colonoscopy

Exclusion Criteria:

* Illiteracy in Dutch and audiovisual or mental handicaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bowel Cleanliness during colonoscopy measured with the Boston Bowel Preparation Scale | During colonoscopy
  Bowel Cleanliness during colonoscopy measured by the endoscopist. The tool used was the Boston Bowel Preparation Scale (Cumulative score of three bowel segments, graded 0-3. Total 10-point scale, ranging from 0=unsatisfactory, 9=excellent).
Bowel Cleanliness during colonoscopy measured with the Ottowa Bowel Preparation Scale | During colonoscopy
  Bowel Cleanliness during colonoscopy measured by the endoscopist. The tool used was the Ottowa Bowel Preparation Scale (Cumulative score of three bowel segments, 0 is excellent, 4 is poor. Two points can be added for fluid residue in the complete colon. Total 14-point scale, ranging from 14=completely unprepared, 0=perfect).

SECONDARY OUTCOMES:
Patient Comfort was measured in a five-point Likert scale | Multiple time points: in the hour after instruction, one hour before colonoscopy and two hours after colonoscopy
  Comfort regarding the colonoscopy was measured in a five-point Likert scale ("How comfortable are you") after the moment of informing (nurse and CAI), prior to colonoscopy and after colonoscopy
Anxiety was measured in a five-point Likert scale | Multiple time points: in the hour after instruction and one hour before colonoscopy
  Anxiety regarding the colonoscopy was measured in a five-point Likert scale ("How anxious are you") after the moment of informing (nurse and CAI) and prior to colonoscopy.
Knowledge and comprehension prior to colonoscopy was measured in a 10 questions knowledge test | One hour before colonoscopy
  Comprehension before colonoscopy was measured in a 10 questions knowledge test on information prior provided.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Klemt-Kropp, MD PhD, Principal Investigator — Medical Centre Alkmaar

IPD SHARING:
Plan to Share IPD: No